CLINICAL TRIAL: NCT01348997
Title: E-Health Intervention for Cancer Survivors 2.0
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study ended prior to completion of planning stage. No participants enrolled.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU Lurie 10CC01
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Cancer
Keywords: cancer; cancer survivors; internet; depression; anxiety
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project Onward website + 16 person social network (Active Comparator)
  Interventions: Behavioral: Project Onward website + 16 person social network
- Project Onward website + 8 person social network (Active Comparator)
  Interventions: Behavioral: Project Onward website + 8 person social network

INTERVENTIONS:
Behavioral: Project Onward website + 16 person social network — The website will include 8 weeks of Internet-based cognitive behavioral therapy combined with discussion and support from a group of up to 16 other cancer survivors.
  Arms: Project Onward website + 16 person social network
Behavioral: Project Onward website + 8 person social network — The website will include 8 weeks of Internet-based cognitive behavioral therapy combined with discussion and support from a group of up to 8 other cancer survivors.
  Arms: Project Onward website + 8 person social network

SUMMARY:
This study will develop and examine the effectiveness of an intervention that utilizes technology to improve cancer survivors' access to mental health care and increase their ability to manage the stressors involved in cancer survivorship. The intervention, referred to as Project Onward, uses an interactive website and an online social network. The purpose of this study is to pilot a novel intervention that can reduce costs, examine methods to improve adherence to internet based treatment and overcome numerous barriers to treatment for mental health concerns.

DETAILED DESCRIPTION:
Nearly 65% of those with cancer diagnoses will survive for at least 5 years, with approximately 10.5 million cancer survivors in the United States. The time of transition for cancer patients, from active treatment to survivorship, has been identified as a time of high risk for depression and anxiety. Cancer survivors experience higher rates of anxiety and depression than those without a cancer history. Research has identified fear of recurrence, perceived loss of support, and social pressure to resume a "normal" life, among other phenomena, as sources for this emotional distress. However, only about 20% of all patients referred for psychotherapy ever enter treatment and of those who initiate treatment, nearly half drop out before completion. This suggests that there are significant barriers to receiving care. These barriers may be even higher for cancer survivors struggling with issues related to re-entry, such as returning to work, resuming household responsibilities and managing residual symptoms such as fatigue or pain.

The internet promises to provide inexpensive access to treatment at any time of the day or night. Unfortunately, the potential for internet delivered services has not been realized. Studies examining treatments that simply provide access to an internet site commonly result in very high dropout after the first site visit, and typically little or no improvement target symptoms. A variety of methods to improve responses to internet interventions have been examined. In general, e-mail support improves adherence and telephone support can improve adherence even more. Another type of support that has only begun to be investigated is the use of social networks to help maintain adherence.

This intervention will use an online social network, to increase adherence and promote the use of the website and the skills it teaches.

ELIGIBILITY:
Inclusion Criteria:

* Any cancer diagnosis.
* Has completed treatment for cancer and is currently in full remission.
* ECOG performance Status of < 3.
* Has a telephone, e-mail account, computer, and broadband access to the Internet.
* Has familiarity with using the Internet that allows for adequate navigation of website.
* Is able to speak and read English.
* Is at least 19 years of age.
* Is able to give informed consent.

Exclusion Criteria:

* Has visual impairment that would prevent use of the website and completion of assessment materials.
* Diagnosis of basal or squamous cell skin cancers.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Depression, as measured by the Hospital Anxiety and Depression Scale (HADS) | Measured at baseline, 4 weeks, 8 weeks and 12 weeks
Anxiety, as measured by the Hospital Anxiety and Depression Scale (HADS) | Measured at baseline, 4 weeks, 8 weeks and 12 weeks

SECONDARY OUTCOMES:
Website utilization (e.g., number of logins, average visit length, total time spent on the site, number of exercises completed) | From baseline through 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mohr, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States